CLINICAL TRIAL: NCT01696955
Title: A Randomized Phase II Trial of ARQ 197 (Tivantinib)/Cetuximab Versus Cetuximab in Patients With Recurrent/Metastatic Head and Neck Cancer
Brief Title: Cetuximab With or Without Tivantinib in Treating Patients With Head and Neck Cancer That Is Recurrent, Metastatic, or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01640; NCI-2012-01640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-1359; 478834; 9165 (Other: University of Chicago Comprehensive Cancer Center); 9165 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (cetuximab and tivantinib) (Experimental): Patients receive cetuximab IV over 60-120 minutes on days 1 and 15 and tivantinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Other: Laboratory Biomarker Analysis; Drug: Tivantinib
- Arm II (cetuximab) (Experimental): Patients receive cetuximab IV over 60-120 minutes on days 1 and 15. Patients who fail cetuximab as a single agent may receive single agent tivantinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Cetuximab — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tivantinib — Given PO
  Arms: Arm I (cetuximab and tivantinib)

SUMMARY:
This randomized phase II trial studies how well cetuximab with or without tivantinib works in treating patients with head and neck cancer that has come back (recurrent), has spread to other places in the body (metastatic), or cannot be removed by surgery. Monoclonal antibodies, such as cetuximab, may interfere with the ability of tumor cells to grow and spread. Tivantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether cetuximab is more effective with or without tivantinib in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Response rate (comparing the cetuximab/ARQ 197 [tivantinib] combination with cetuximab single agent activity).

SECONDARY OBJECTIVES:

I. Continuous tumor shrinkage. II. Progression-free survival (PFS). III. Overall survival (OS). IV. Objectives I, II, and III above, as well as response rates, will be assessed and compared between treatment arms in the subgroup of patients with high mesenchymal epithelial transition factor (c-MET) expression, and/or high c-MET copy number.

V. Single agent activity for ARQ 197 (tivantinib) in patients who have failed cetuximab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cetuximab intravenously (IV) over 60-120 minutes on days 1 and 15 and tivantinib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cetuximab IV over 60-120 minutes on days 1 and 15. Patients who fail cetuximab as a single agent may receive single agent tivantinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of squamous cell carcinoma of head and neck origin not amenable to curative intent therapy; both human papillomavirus (HPV) positive (+) and HPV negative (-) are eligible, but status has to be known prior to randomization (although not required for consenting); any type of tissue based HPV assessment is acceptable (e.g. p16 immunohistochemistry [IHC] or HPV in situ hybridization [ISH]); if local HPV testing is not available slides can be sent to the University of Chicago for HPV testing; please note that p16 IHC is generally only considered to be accurate for oropharyngeal tumors
* Presence of measurable lesions (as per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1); generally a >= 10 mm tumor lesion (in the longest diameter by computed tomography [CT] scan) or a lymph node >= 15 mm (short axis) is considered measurable disease when evaluated by CT scan (with a slice thickness no greater than 5 mm)
* Availability of tissue (10 tumor containing formalin-fixed, paraffin-embedded [FFPE] slides/sections)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1
* Patients who have received cetuximab or another inhibitor of epidermal growth factor receptor (EGFR) in the curative intent treatment setting (e.g. with radiation or during induction chemotherapy [prior to definitive, curative intent therapy]) are eligible for the study
* Life expectancy of greater than 8 weeks
* Hemoglobin >= 9.0 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must be able to swallow ARQ 197 (tivantinib) by mouth, unless adequate data about administration by gastrostomy (G)-tube becomes available; tablets may be crushed, but must be taken orally
* Human immunodeficiency virus (HIV)-positive patients with normal immune function (cluster of differentiation [CD]4 count > 200) are eligible if there are no drug interactions with ARQ 197 (tivantinib) or cetuximab
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ARQ 197 (tivantinib) administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Nasopharyngeal tumors that show lymphoepithelioma histology
* Patients who have received more than 2 prior cytotoxic treatments in the palliative treatment setting are ineligible
* Patients who have received treatment with an EGFR or MET inhibitor in the palliative treatment setting are ineligible
* Patients with known, active brain metastases should be excluded from this clinical trial; patients with treated brain metastases stable for >= 12 weeks are eligible; use of corticosteroid (for patients with brain metastasis and other indications for corticosteroid use) is acceptable on a low maintenance or tapering dose schedule
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ARQ 197 (tivantinib) or cetuximab
* Concurrent life-threatening diseases: patients with diseases which with reasonable certainty do not limit life expectancy to 12 months or less are eligible; assessment of such concurrent illnesses should be by the principal investigator
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ARQ 197 (tivantinib)
* Concurrent use of warfarin (therapeutic use) is allowed, but requires close monitoring of prothrombin time (PT)/international normalized ratio (INR)
* History of congestive heart failure defined as class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD), clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as >= grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Patients may not be receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (24):
- United States (24):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Cetuximab and Tivantinib): Patients receive cetuximab 500mg/m2 IV over 60-120 minutes on days 1 and 15 and tivantinib 360mg PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cetuximab: Given IV
  Tivantinib: Given PO
- Arm II (Cetuximab): Patients receive cetuximab 500 mg/m2 IV over 60-120 minutes on days 1 and 15. Patients who fail (progress) on cetuximab as a single agent may then receive single agent tivantinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cetuximab: Given IV
Period: Main Study
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Started | 42 | 39
Completed | 40 | 38
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Failure on Cetuximab-Received Tivantinib
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Started | 0 | 15
Completed | 0 | 15 (23 patients did not cross over)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm II (Cetuximab): Patients receive cetuximab 500mg/m2 IV over 60-120 minutes on days 1 and 15. Patients who fail (progress) on cetuximab as a single agent may then receive single agent tivantinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cetuximab: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab) | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [37 to 90] | 63.6 [35 to 87] | 62.0 [35 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 34 | 32 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 32 | 33 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 40 | 38
Participants
  Complete response | 1 | 0
  Partial response | 2 | 3
Statistical Analysis 1: Comparison: Arm I (Cetuximab and Tivantinib) vs Arm II (Cetuximab); Test type: Superiority; p = 0.99, Fisher Exact

2. Secondary Outcome: c-MET Copy Number
Description: Change in copy number from baseline to 8 weeks
Time Frame: Baseline to 8 weeks
Population: Assay not performed.
Groups:
- Arm I (Cetuximab and Tivantinib): Patients receive cetuximab 500 mg/m2 IV over 60-120 minutes on days 1 and 15 and tivantinib 360 mg PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cetuximab: Given IV
  Tivantinib: Given PO
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: c-MET Expression
Description: Change in c-MET expression from baseline to 8 weeks
Time Frame: Baseline to 8 weeks
Population: Assay not performed.
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Tumor Burden
Description: Early change in tumor burden measured using the sum of longest diameters of target lesions, expressed as percent change from baseline.
Time Frame: Baseline to 8 weeks
Population: Patients with baseline and 8 week measurements available
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Arm I (Cetuximab and Tivantinib): Patients receive cetuximab 500 mg/m2 IV over 60-120 minutes on days 1 and 15 and tivantinib 360mg PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Cetuximab: Given IV
  Tivantinib: Given PO
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 32 | 31
percent change | 15.0 (6.1) | 9.0 (5.5)
Statistical Analysis 1: Comparison: Arm I (Cetuximab and Tivantinib) vs Arm II (Cetuximab); Test type: Superiority; p = 0.47, t-test, 2 sided

5. Secondary Outcome: Overall Survival
Description: Time from randomization until death or date last known alive
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 40 | 38
months | 7.4 [4.7 to 10.3] | 8.6 [5.7 to 11.5]
Statistical Analysis 1: Comparison: Arm I (Cetuximab and Tivantinib) vs Arm II (Cetuximab); Test type: Superiority; p = 0.99, Log Rank

6. Secondary Outcome: Progression-free Survival
Description: Time from randomization until disease progression/death from any cause or date last know progression-free
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab)
Number analyzed (Participants) | 40 | 38
months | 3.5 [1.8 to 3.9] | 3.5 [2.0 to 3.9]
Statistical Analysis 1: Comparison: Arm I (Cetuximab and Tivantinib) vs Arm II (Cetuximab); Test type: Superiority; p = 0.58, Log Rank

7. Secondary Outcome: Overall Response Rate of Single-agent Tivantinib After Failure of Cetuximab
Description: as for outcome 1
Time Frame: Up to 1 year
Population: This outcome pertains only to Tivantinib after Cetuximab failure and therefore Arm 1 contains 0 analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Tivantinib After Cetuximab Failure: ARQ 197 (tivantinib) 360mg PO BID on days 1-28.
Arm/Group | Arm I (Cetuximab and Tivantinib) | Tivantinib After Cetuximab Failure
Number analyzed (Participants) | 0 | 15
Participants |  | 0

8. Other Pre Specified Outcome: Number of Participants With Adverse Events While on Single-agent Tivantinib After Failure of Cetuximab
Description: Non-serious adverse events, CTCAE (4.0)
Time Frame: Up to 3 years
Population: This outcome pertains only to Tivantinib after Cetuximab Failure and therefore Arm 1 contains 0 analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab and Tivantinib) | Tivantinib After Cetuximab Failure
Number analyzed (Participants) | 0 | 15
Participants |  | 9

9. Other Pre Specified Outcome: Number of Patients With Serious Adverse Events While on Single-agent Tivantinib After Failure of Cetuximab
Description: CTCAE (4.0)
Time Frame: 3 years
Population: This outcome pertains only to Tivantinib after Cetuximab Failure and therefore Arm 1 contains 0 analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cetuximab and Tivantinib) | Tivantinib After Cetuximab Failure
Number analyzed (Participants) | 0 | 15
Participants |  | 4

ADVERSE EVENTS:
Time Frame: 3 years
Description: Note: Adverse events reported in Arm II were prior to any crossover to combination therapy.
Groups:
- Single-agent Tivantinib After Failure of Cetuximab: Patients receive cetuximab 500mg/m2 IV over 60-120 minutes on days 1 and 15.
Arm/Group | Arm I (Cetuximab and Tivantinib) | Arm II (Cetuximab) | Single-agent Tivantinib After Failure of Cetuximab
All-Cause Mortality (participants affected / at risk) | 36/40 | 35/38 | 2/15
Serious Adverse Events (participants affected / at risk) | 19/40 | 18/38 | 4/15
Other Adverse Events (participants affected / at risk) | 38/40 | 35/38 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cetuximab and Tivantinib) (N=40) | Arm II (Cetuximab) (N=38) | Single-agent Tivantinib After Failure of Cetuximab (N=15)
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1
Cardiac arrest (Investigations) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Death NOS (General disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Fever (General disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 1 | 0 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tracheal hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
White blood cell decreased (Investigations) | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 1
Infections - Other (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cetuximab and Tivantinib) (N=40) | Arm II (Cetuximab) (N=38) | Single-agent Tivantinib After Failure of Cetuximab (N=15)
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0
Alkaline phosphatase increased (Investigations) | 6 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 16 | 9 | 3
Anorexia (Metabolism and nutrition disorders) | 12 | 10 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Blood bilirubin increased (Investigations) | 3 | 2 | 0
Chills (General disorders) | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 10 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 2
Dysgeusia (Nervous system disorders) | 3 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Edema limbs (General disorders) | 5 | 1 | 1
Fatigue (General disorders) | 21 | 17 | 3
Headache (Nervous system disorders) | 3 | 5 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypertension (Vascular disorders) | 5 | 5 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 6 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 6 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 10 | 3
Hyponatremia (Metabolism and nutrition disorders) | 11 | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 5 | 2
Infusion related reaction (General disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 10 | 4 | 3
Nausea (Gastrointestinal disorders) | 12 | 10 | 1
Neutrophil count decreased (Investigations) | 8 | 1 | 0
Platelet count decreased (Investigations) | 9 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 20 | 19 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 10 | 2
Rash/dermatitis (Skin and subcutaneous tissue disorders) | 6 | 8 | 1
Sinus bradycardia (Cardiac disorders) | 8 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
Pharyngitis (Infections and infestations) | 10 | 6 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6 | 1
White blood cell decreased (Investigations) | 9 | 6 | 1
Anxiety (Psychiatric disorders) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Creatinine increased (Investigations) | 0 | 3 | 1
Edema face (General disorders) | 1 | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fever (General disorders) | 2 | 4 | 1
Flu like symptoms (Gastrointestinal disorders) | 0 | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 2
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Oral pain (Gastrointestinal disorders) | 2 | 3 | 0
Pain (General disorders) | 2 | 3 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT01696955/Prot_SAP_000.pdf